CLINICAL TRIAL: NCT01920243
Title: Applying Health Mechanics to Enhance Bowel and Bladder Health for Persons With SCI
Brief Title: Evaluation of a Bowel and Bladder Health Management Program for Individuals With Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle Meade, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H133N110002 -2
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Injuries, Spinal Cord; Neurogenic Bowel; Urinary Bladder, Neurogenic
Keywords: Telemedicine; self-management; Medical psychology; Health psychology; Rehabilitation; Education, Health
MeSH Terms: conditions — Spinal Cord Injuries; Neurogenic Bowel; Urinary Bladder, Neurogenic; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Health Mechanics- New Injuries (Experimental): The Health Mechanics Program group receives the intervention. For this study, the Health Mechanics protocol is being applied to two areas of SCI management, bladder and bowel management, and administered over the telephone. The intervention will be administered as a series of modules delivered by a Health Coach (a health professional who works within the study team and is knowledgeable about SCI management). Individuals with new-onset traumatic spinal cord injuries are eligible for this group.
  Interventions: Behavioral: Health Mechanics Program
- Usual Care- New Injuries (No Intervention): This group will not receive the intervention. They will receive usual care. This group will be comprised of individuals with new-onset traumatic spinal cord injuries.
- Health Mechanics- Chronic Injuries (Experimental): The Health Mechanics Program group receives the intervention. For this study, the Health Mechanics protocol is being applied to two areas of SCI management, bladder and bowel management, and administered over the telephone. The intervention will be administered as a series of modules delivered by a Health Coach (a health professional who works within the study team and is knowledgeable about SCI management). Individuals who have had traumatic spinal cord injuries for at least one year are eligible for this group.
  Interventions: Behavioral: Health Mechanics Program
- Usual Care- Chronics (No Intervention): This group will not receive the intervention. They will receive usual care. This group will be comprised of individuals with who have had traumatic spinal cord injuries for at least one year.

INTERVENTIONS:
Behavioral: Health Mechanics Program — The intervention will consist of six modules that will address attitudes, self-monitoring, communication and organizational skills, problem solving skills and stress management as presented through the Health Mechanics program. These modules are designed to take place over 6 phone calls of approximately 45 minutes each. In order to provide flexibility for the participants, the quantity and duration of calls may vary depending on the extent that the participant completes the homework and the amount of time they need to learn the skill.
  Other Names: Health Mechanics
  Arms: Health Mechanics- Chronic Injuries; Health Mechanics- New Injuries

SUMMARY:
This study will look at the use of a telehealth version of a self management program in individuals with both new onset and chronic traumatic spinal cord injuries. The program is called Health Mechanics. It is meant to enhance self management skills related to neurogenic bladder and bowel management to prevent associated problems and improve Quality of Life (QOL). This program is based on the needs and strengths of individuals with SCI. It focuses on enhancing skills, encouraging positive health behaviors, empowering people within their own environments, and recognizing that people differ in their resources and abilities. The skills that are part of the intervention are: attitude, self-monitoring, problem-solving, communication, organization and stress management. This study will address those skills in the context of bladder and bowel health, with expectations that these skills to be useful in other areas of life as well.

The investigators hypothesize that individuals in the Health Mechanics intervention group will:

* show greater improvements in problem solving skills, healthy attitudes about disability and knowledge of SCI management skills than will the control group
* have greater adherence to recommended bladder and bowel management behaviors than the control group
* have fewer bladder and bowel complications than the control group
* have higher levels of QOL than the control group

In other words, this study will investigate the effectiveness of a telehealth version of Health Mechanics to enhance self-management skills related to neurogenic bladder and bowel management in an attempt to prevent associated complications and improve QOL.

DETAILED DESCRIPTION:
Background and Overview

This study will evaluate the efficacy of a newly developed self-management program, Health Mechanics, to develop and improve bladder and bowel management skills among persons with new and chronic SCI. Program participation is expected to prevent bladder and bowel related medical complications (e.g., constipation, leakage), leading to enhanced social participation and QOL. Health Mechanics was designed by the study PI, Dr. Meade, between 2007 and 2009 with funding from the Paralyzed Veteran's of America Education Foundation to assist persons with SCI develop and transfer the necessary skills to keep their bodies healthy while managing the many aspects of SCI care.

This study will investigate the effectiveness of a telehealth version of Health Mechanics to enhance self-management skills related to neurogenic bladder and bowel management in an attempt to prevent associated complications and improve QOL. The study makes a unique contribution to rehabilitation by emphasizing the concepts of personal responsibility and control over one's health and life as a whole. By selecting a telehealth approach (here defined as telephone-based) for program implementation, the investigators also attempt to address the high cost of care delivery and lack of health care access to underserved populations with SCI living in remote areas of the State of Michigan.

The Health Mechanics program is designed based on the needs and strengths of individuals with SCI while being responsive to identified gaps and challenges of health care provision in this population. The program focuses on enhancing skills, encouraging positive health behaviors and empowering people within their own environments, recognizing that people have different resources and abilities. For this study, the Health Mechanics program has been adapted to specifically focus on bladder and bowel management related concerns and to be administered via telephone, thus better addressing the needs of the rural population and transportation-related challenges.

By teaching skills to better manage bladder and bowel health, this self-management program should not only reduce the occurrence of complications but it should also result in higher levels of social integration and QOL. Since the skills taught - attitude, self-monitoring, problem-solving, communication, organization and stress management - will be addressed in the context of performing the behaviors necessary to enhance bladder and bowel health, we expect them to generalize into other areas such that improvements in these skills result in better overall health and participation.

Purpose and Objectives

The proposed study's overall purpose is to evaluate the effects of Health Mechanics in preventing bladder and bowel complications and to improve QOL. The program specifically targets newly injured individuals for early prevention of complications, as well individuals with chronic injuries for later treatment and prevention of complications. Objectives are: 1) to improve self-management skills, including problem-solving, knowledge of health behaviors, and attitude about disability; 2) to increase adherence to recommended bladder and bowel management behaviors; 3) to improve bladder and bowel health and related QOL; and 4) to determine the extent that program improvements in terms of skills acquired are sustained over time. Short-term refers to 3 and 6 months assessments while long-term refers to the 12 month assessment. All hypotheses posit that, following the intervention, differences will exist such that participants in the Health Mechanics program will perform better than the control group (an assessment of between group differences) and that these differences will be sustained over time (an assessment of within and between group differences). It is expected that individuals with new injuries will improve over time regardless of group assignment, while individuals with chronic injuries are stabilized prior to admission to the study. Because of these naturally occurring differences in trajectory, we will be examining within and between group differences.

Research Hypotheses

H1: Program participants will show greater improvements in problem solving skills, healthy attitudes about disability and knowledge of SCI management skills than will the control group; these improvements will be sustained over time within and between groups.

H2: Program participants will have greater adherence to recommended bladder and bowel management behaviors than the control group; these improvements will be sustained over time within and between groups.

H3: Program participants will have fewer bladder and bowel complications than the members of the control group; these differences will be maintained over time within and between groups.

H4: Program participants will have higher levels of QOL than the control group; these differences will be sustained over time within and between groups.

ELIGIBILITY:
Inclusion Criteria for all groups:

* having a traumatic spinal cord injury
* being at least 18 years old
* having neurogenic bowel and/or bladder
* being community-living
* English-speaking

Additional inclusion criteria for new injury onset groups:

* completing inpatient rehabilitation for new SCI at University of Michigan Health System

Additional inclusion criteria for chronic injury groups:

* having an SCI for at least one year before enrollment
* expressing moderate to occasional bowel and/or bladder issues on the secondary conditions scale with associated distress

Exclusion Criteria for all groups:

* cognitive deficits and psychiatric conditions that render persons unable to independently direct or perform their own care

Additional Exclusion Criteria for chronic injury groups:

* current episode of severe depression as evidenced by scoring 20 or higher on the PHQ-9
* current suicidality or suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Spinal Cord Injury Quality of Life (SCI-QOL) Emotional Domain | Change from baseline at 6-month assessment
  The SCIQOL is administered via computerized adaptive testing forms and measures specific domains of health related quality of life relevant to living with SCI.
SCI-QOL Physical Domain | Change from baseline at 6-month assessment
  The SCIQOL is administered via computerized adaptive testing forms and measures specific domains of health related quality of life relevant to living with SCI.
SCI-QOL Social Domain | 6-month assessment
  The SCIQOL is administered via computerized adaptive testing forms and measures specific domains of health related quality of life relevant to living with SCI. This outcome will measure between group differences.
Bowel and Bladder Treatment Index (BBTI) | Change from baseline at 6-month assessment
  The BBTI is a means for identification of the main method used for defecation as well as bladder management. It also measures complications and overall bowel and bladder health.

SECONDARY OUTCOMES:
Adapted version of the SCI Knowledge Questionnaire - SF | Change from baseline at 6-month assessment
  Adapted from Thietje et al. (2011) this measure assesses knowledge of bladder and bowel management
Social Problem Solving Inventory - Revised: Short Form (SPSI-R:S) | Change from baseline at 6-month assessment
  Measures four dimensions of problem solving: negative problem orientation, rational problem solving, impulsivity/carelessness and avoidance.
Appraisals of Disability: Primary and Secondary Scale (ADAPSS) | Change from baseline at 6-month assessment
  Measures six dimensions of appraisal: fearful despondency, overwhelming disbelief, determined resolve, growth and resilience, negative perceptions of disability, and personal agency.
Disability Management Self Efficacy Scale (DMSES) - SF | Change from baseline at 6-month assessment
  Measures perceived ability to manage SCI related tasks
Behavioral Adherence Assessment of Bladder and Bowel Treatment (BAABBT) | Change from baseline at 6-month assessment
  The difference between prescribed (by physician) and actual behaviors related specifically to bladder and bowel methods of management
The Craig Handicap Assessment and Reporting Technique, Short Form (CHART-SF) | 6-month assessment
  Assessment of time spent performing a variety of activities in the home and community. This outcome will measure between group differences.

OTHER OUTCOMES:
Process Evaluation | 6-month assessment
  Provides an opportunity for the participant to inform the research study team on his/her experience with the intervention and assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Meade, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Spinal Cord Injury Model System, Ann Arbor, Michigan, United States